CLINICAL TRIAL: NCT04807842
Title: A Double-blind, Randomized, Placebo-controlled Study to Confirm the Efficacy and Safety of Multi- Gyn ActiGel Plus for Treatment of Bacterial Vaginosis
Brief Title: Multi-Gyn ActiGel Plus for Treatment of Bacterial Vaginosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioClin BV (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Organization: Karo Pharma AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGAP BV 001
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-03

CONDITIONS: Bacterial Vaginoses
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: double blinded, randomized placebo controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active product (Other)
  Interventions: Device: vaginal gel
- Placebo (Placebo Comparator)
  Interventions: Device: vaginal gel

INTERVENTIONS:
Device: vaginal gel — The placebo gel is a non-buffered gel. The active device is an acidic gel.

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical investigation. The objective of the study is to confirm the efficacy of Multi-Gyn ActiGel Plus to treat BV as compared to a placebo control.

Treatment arm 1: Multi-Gyn ActiGel Plus Treatment arm 2: placebo gel Both the Multi-Gyn ActiGel Plus and the placebo will be applied twice a day for 7 consecutive days. Visit 2 will be performed at 3 weeks after start of treatment A phone call will take place, at 5 weeks after start of treatment for subject with clinical cure at Visit 2. The total duration per subject is estimated 5 weeks and the total study duration is 13 months. Sample size is 100 subjects per treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with BV (3 out of 4 Amsel criteria positive, with at least presence of clue cells (>20%))
* Women of childbearing potential
* Aged >18 years
* Signed written informed consent form
* Willing to comply to the follow-up schedule

Exclusion Criteria:

* Current clinically manifest of sexually transmitted gynecologically infection, genital tract infection, vulvovaginal candidosis or aerobic vaginitis (incl. clinical obvious gonorrhoea, chlamydia trachomatis or mycoplasma genitalium infection with cervicitis, urethritis, salpingitis)
* Presence of Trichomonas and/or Candida Albicans in vaginal smear during examination of the smears for Amstel criteria (clue cells detection)
* Current genital malignancies
* Chemotherapy for any reason in last 6 months
* Radiotherapy in the genitourinary system in the last 12 months
* Use of antibiotics for any reason in the last 14 days
* Use of intravaginal devices during the investigation or in the last 14 days
* Pregnancy or currently attempting to conceive
* Lactation
* Use of other treatment for vaginal conditions during the course of the clinical investigation
* Known allergies to ingredients of the product
* Concomitant medication for treatment of vaginal infections, or other use of intravaginal medication during the course of the clinical investigation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate of BV at 3 weeks after start of treatment (end-of treatment visit; Visit 2). | 3 weeks
  Clinical cure is defined based on the following Amsel criteria:
  1. presence of clue cells <20% of the total epithelial cells on microscopic examination of the saline wet mount
  2. resolution of the abnormal vaginal discharge, and
  3. a negative whiff test

SECONDARY OUTCOMES:
Microbiological cure rate (based on Nugent score <4) at Visit 2 | 3 weeks
  The secondary objective of the study is to confirm the secondary efficacy of the product.

CONTACTS AND LOCATIONS:
Locations (1):
- Praxis Dr. Peters, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No